CLINICAL TRIAL: NCT04577742
Title: Long-term Outcomes in Uveal Melanoma After Ruthenium-106 Brachytherapy
Brief Title: Uveal Melanoma and Brachytheraphy: Long-term Outcomes.
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 2020/106
Record Dates: First submitted 2020-10-03; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: 106 Ruthenium Plaque Brachytherapy; Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: 106 Ruthenium plaque brachytherapy — All patients, affected by uveal melanoma, were treated with 106 Ruthenium plaque brachytherapy to a total dose of 100 Gy to the tumor apex. The time of implant duration was calculated according to the conventional central-axis-point dose calculation

SUMMARY:
This study investigated the visual and anatomical outcomes, tumor control, tumor recurrence, distant metastasis and cancer free survival in patients affected by uveal melanoma and undergoing Ru-106 plaque brachytherapy between February 2011 and March 2020

ELIGIBILITY:
Inclusion Criteria:

* age older than 40 years
* diagnosis of uveal melanoma

Exclusion Criteria:

* age older than 80 years
* No diagnosis of uveal melanoma

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participans were older than 40 years with uveal melanoma and they underwent Ruthenium 106 brachytherapy
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
To evaluate long-term outcomes in patients underwent brachytherapy for uveal melanoma | Mean follow-up was 4 years (3 months-9 years)
  To investigate the visual and anatomical outcomes, tumor control, tumor recurrence, distant metastasis and cancer free survival

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II", Naples, Italy